CLINICAL TRIAL: NCT04398797
Title: Prevention of AcuTe admIssioN Algorithm (PATINA) - The Effect of a Notification Algorithm and a Digital Decision Support Tool
Brief Title: Prevention of AcuTe admIssioN Algorithm (PATINA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region of Southern Denmark (Other)
Collaborators: Odense Municipality, Denmark (Unknown); Kerteminde Municipality, Denmark (Unknown); Svendborg Municipality, Denmark (Unknown)
Responsible Party: Principal Investigator, Anders Fournaise, Industrial PhD student, Region of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19/29873; 9163-00002B (Other Grant/Funding Number: Innovation Fund Denmark); 19/20991 (Other Grant/Funding Number: Region of Southern Denmark); OP_1033 (Other: Open Patient data Explorative Network (OPEN))
Record Dates: First submitted 2020-05-13; First posted 2020-05-21 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Avoid Acute Hospitalizations
Keywords: Algorithm; Community dwelling; Health care utilization; Acute hospitalization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Step-wedge, open label, cluster randomized controlled trial with 1 year follow up. Area home care teams from three Danish municipalities are randomized to cross-over from the control phase to the intervention phase. Participants automatically follow their area home care team into the allocated group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Use of notification algorithm and nurse follow-up
  Interventions: Other: PATINA algorithm
- Control (No Intervention): Standard regime (usual care)

INTERVENTIONS:
Other: PATINA algorithm — Once a week community nurses receive a list of community dwelling citizens deemed at risk of deterioration that can lead to hospital admission. Nurses assess each citizens situation and initiate intervention if needed (not part of the intervention).
  Arms: Intervention

SUMMARY:
Utilization of public health care mirrors the older individual's overall health, and increased need for health care may precede more clear symptoms of acute disease. In a previous retrospective study, we found a significant increase in municipal home care service (minutes/week) in a 12-month period prior to acute hospitalization. This PhD-study aims at examining the effect of a software algorithm monitoring older citizens utilization of municipal home care. When home care increases the community nurse is notified and special attention is paid to the individual's current health situation. Pro-active health care initiatives may be launched in collaboration with the primary care physician. The intervention is the algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling citizens (+ 65) receiving home and social care in Odense, Kerteminde and Svendborg Municipalities.

Exclusion Criteria:

* Non

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2464 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Hospitalizations | 30 days from identification by the algorithm (6 months for intervention phase)
  Calculated based on data from the Danish National Patient Registry

SECONDARY OUTCOMES:
Hospital readmissions | 30 days from identification by the algorithm (6 months for intervention phase)
  Calculated based on data from the Danish National Patient Registry
Outpatient contacts | 30 days from identification by the algorithm (6 months for intervention phase)
  Calculated based on data from the Danish National Patient Registry
Use of temporary care in a skilled nursing facility | 30 days from identification by the algorithm (6 months for intervention phase)
  Calculated based on data from the three participating municipalities electronic care records
Use of community home and social care services | 30 days from identification by the algorithm (6 months for intervention phase)
  Calculated based on data from the three participating municipalities electronic care records
Contacts to primary care physicians | 30 days from identification by the algorithm (6 months for intervention phase)
  Calculated based on data from the Danish National Health Insurance Service Register
Mortality | 30 days from identification by the algorithm (6 months for intervention phase)
  Calculated based on data from the Danish Cause of death register.

OTHER OUTCOMES:
Barriers and facilitators for nurse's acceptance of using the algorithm | 30 days from identification by the algorithm (6 months for intervention phase)
  Calculated based on a survey battery collected 1 month pre intervention start, 14-7 days pre intervention start, 1 month post intervention start
Health economic analysis | 1 year
  The analytic details will be based on the primary and secondary results of the trail

CONTACTS AND LOCATIONS:
Overall Officials: Anders Fournaise, MSPH, Principal Investigator — Region of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fournaise A, Lauridsen JT, Bech M, Wiil UK, Rasmussen JB, Kidholm K, Espersen K, Andersen-Ranberg K. Prevention of AcuTe admIssioN algorithm (PATINA): study protocol of a stepped wedge randomized controlled trial. BMC Geriatr. 2021 Feb 27;21(1):146. doi: 10.1186/s12877-021-02092-2. PMID 33639833